CLINICAL TRIAL: NCT01646515
Title: Udenafil Therapy to Improve Symptomatology, Exercise Tolerance and Hemodynamics in Patients With Chronic Systolic Heart Failure
Acronym: ULTIMATE-SHF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Substantial benefit was observed in the active treatment group
Sponsor: Seoul National University Hospital (Other)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Hyung-Kwan Kim, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-1102-063-352
Record Dates: First submitted 2012-06-13; First posted 2012-07-20 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Systolic Heart Failure
Keywords: systolic heart failure; udenafil; exercise capacity
MeSH Terms: conditions — Heart Failure, Systolic | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo arm (Placebo Comparator): Capsule that is identically appearing with udenafil will be administered to patients in placebo group. For the first 4 weeks, patients will receive 50 mg of placebo drug two times a day, and then the dosage will be doubled to 100 mg two times a day for next 8 weeks.
  Interventions: Drug: Placebo
- Udenafil (Active Comparator): Patients will receive 50 mg of udenafil two times a day, and then the dosage will be doubled to 100 mg two times a day for next 8 weeks.
  Interventions: Drug: Udenafil (Zydena)

INTERVENTIONS:
Drug: Placebo — Capsule, appears identical with udenafil, will be provided by Dong-A pharmaceutical company.
  Patients will receive 50 mg of placebo drug two times a day for 4 weeks, and then the dosage will be escalated to 100 mg two times a day for next 8 weeks
  Arms: placebo arm
Drug: Udenafil (Zydena) — Udenafil (Zydena), a newly developed PDE-5 inhibitor by Dong-A pharmaceutical company, will be administered to patients in this group, 50 mg two times a day for 4 weeks, and then the dosage will be escalated to 100 mg two times a day for next 8 weeks.
  Arms: Udenafil

SUMMARY:
The purpose of this study is to determine if udenafil improves exercise tolerance in patients with systolic heart failure.

DETAILED DESCRIPTION:
Udenafil (Zydena), a newly developed PDE-5 inhibitor, has been proved to have similar efficacy and safety profile, compared with other PDE-5 inhibitors. Also, laboratory data showed that udenafil inhibits ventricular hypertrophy and fibrosis in rat heart failure model. Based on these results, the investigators hypothesized that udenafil would improve symptom, exercise capacity and hemodynamic status in patients with systolic heart failure. In this 12-week, randomized, double-blind, placebo-controlled trial, patients with systolic heart failure will be enrolled according to the eligibility criteria. After randomization, study participants will be assigned to receive either 50mg of udenafil or placebo two times a day for 4 weeks, and then the dosage will be doubled to 100mg two times a day for next 8 weeks. Participants will attend study visits at baseline and weeks 4 and 12. Physical examination, medical history review, blood sample collection and electrocardiogram will be conducted on each study visits. At baseline and week 12, participants will undergo cardiopulmonary exercise test and exercise echocardiography. At every study visits,researchers will collect health information.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age, LV EF < 40%

Exclusion Criteria:

* long-term use of medications that inhibit cytochrome P450 3A4.
* inability patients with exercise test
* primary pulmonary artery hypertension
* severe hypotension (< 90/50mmHg) or severe hypertension (> 170/100mmHg)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-12; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
VO2max with cardiopulmonary exercise test | Baseline and 12th weeks
  VO2 max was defined as cardiopulmonary exercise capacity
  Comparison between groups and within groups

SECONDARY OUTCOMES:
The changes of left ventricle ejection fraction | baseline and 12 th week
  comparison between groups and within groups
serum BNP level | Baseline, 4th week, and 12th week
  Comparison between groups and within groups
Change of ventilator efficiency (VE/VCO2 slope) in cardiopulmonary exercise test | Baseline and 12th week
  Comparison between groups and within groups
Change of symptomatic status expressed as New York Heart Association (NYHA) functional class | Baseline, 4th week, and 12th week
  Comparison between groups and within groups
Change of pulmonary artery systolic pressure (PASP) in echocardiography at rest and during exercise | Baseline and 12th week
  Comparison between groups and within groups.
Safety endpoint | 12th week
  Safety endpoint during 12 week follow-up, is defined as follows:
  1. Development of facial flushing, febrile sensation, eyeball pain, visual disturbance, headache, penile erection.
  2. Intolerance or development of other adverse drug reactions related with study drug.
Change of symptomatic status expressed as Borg dyspnea index | baseline, 4 weeks and 12 weeks
  Comparison between groups and within groups.

OTHER OUTCOMES:
All cause death, cardiac death, and heart failure-related admission and their composite | 12 week
  All cause death, cardiac death, and heart failure-related admission and their composite

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim KH, Kim HK, Hwang IC, Lee SP, Cho HJ, Kang HJ, Kim YJ, Sohn DW. ULTIMATE-SHF trial (UdenafiL Therapy to Improve symptoMAtology, exercise Tolerance and hEmodynamics in patients with chronic systolic heart failure): study protocol for a randomized, placebo-controlled, double-blind trial. Trials. 2013 Jun 22;14:188. doi: 10.1186/1745-6215-14-188. PMID 23799908